CLINICAL TRIAL: NCT01926574
Title: Evaluation of Inpatient-return- To-work, Multicomponent, Rehabilitation Programs for Persons Temporary Out of Work With Musculoskeletal-, Unspecific-, and/or Common Mental Health Disorders; Randomized Controlled Trial
Brief Title: Evaluation of Return to Work Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2012/1241-1
Record Dates: First submitted 2013-08-19; First posted 2013-08-21 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Sick Leave; Occupational Health
Keywords: absenteeism; rehabilitation; return to work
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- long rehabilitation (Experimental): a 3.5-week, in-patient rehabilitation program, organized as a 7-hour workday with weekends off, simulating a close to normal summer work-week in Norway, and mainly group-based with maximum 8 participants per group. Focus on mental training (aimed at increasing motivation and self-efficacy), physical training and work-related problem solving.
  Interventions: Behavioral: long rehabilitation program
- short rehabilitation (Experimental): 4+4 full days of rehabilitation at Hysnes Rehabilitation Center, separated by 2 weeks living at home. Group-based with 8 participants per group, focus on mental training (aimed at increasing motivation and self-efficacy), physical training and work-related problem solving. A workplace visit will be included in addition to the 4 + 4 rehabilitation days, if considered relevant.
  Interventions: Behavioral: short rehabilitation program
- Acceptance and commitment therapy (Active Comparator): 6 dynamic processes (committed action, self-as-context, presence in the moment, values, defusion and acceptance) are targeted both in group-sessions and individual meetings. Only the psychological part of the experimental interventions is applied, in an outpatient setting.
  Interventions: Behavioral: Acceptance and commitment therapy (ACT)
- Untouched (No Intervention): this group will be followed in registers at group level and not be aware of their participation in the study

INTERVENTIONS:
Behavioral: long rehabilitation program
  Arms: long rehabilitation
Behavioral: short rehabilitation program
  Arms: short rehabilitation
Behavioral: Acceptance and commitment therapy (ACT)
  Arms: Acceptance and commitment therapy

SUMMARY:
Long-term sick-listing from work has considerable impact on social function, on the families of the sick-listed persons, the companies they work for, and society as a whole. Hence, the need for documented effective vocational rehabilitation programs is pressing. Vocational rehabilitation services described in the scientific literature have been specific to one single or a specific group of medical conditions (e.g.low back pain). In contrast, most people on sick leave have several health complaints, and many of the factors influencing sick leave are shared regardless of disorder (e.g. social surroundings, workplace environment), calling for rehabilitation programs that can be employed for both musculoskeletal-, unspecific- and common mental disorders. Aim of this study is to investigate whether a group based rehabilitation program for musculoskeletal, mental or unspecific complaints can facilitate return-to-work (RTW), thereby testing two multicomponent return-to-work RTW rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* living in the counties of Trøndelag
* on sick leave 2-12 months
* current sick leave status of 50% - 100%
* ICPC-2 (International Classification of Primary Care, Second edition) diagnosis within the L (musculoskeletal), P (psychiatric) or A (unspecific disorders) categories

Exclusion Criteria:

* alcohol or drug abuse
* serious somatic or psychological disorders
* a specific disorder requiring specialized treatment
* pregnancy
* currently participating in another treatment program
* insufficient Norwegian speaking or writing skills to participate in group session and fill out questionnaires
* scheduled for surgery within the next 6 months
* serious problems with functioning in a group setting

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
time until full sustainable return-to-work (RTW) | 1 year
  return-to-work i.e. for at least 4 weeks without relapse
Total number of sickness absence days | 1 year
  after enrollment in the study (i.e. after pre-screening)

SECONDARY OUTCOMES:
Sickness absence days | 3 years
sickness absence days | 5 years
Health related quality of life | 1 year
Subjective health complaints | 1 year
  Pain, depression, anxiety, and other subjective complaints
Physical activity | 1 year
physical, social and emotional functional status | 1 year
Psychological and social factors at work | 1 year
readiness for return to work | 1 year
fear avoidance beliefs | 1 year
psychological flexibility and acceptance | 1 year
share of workers at work | 1 year

OTHER OUTCOMES:
Health economics from the societal perspective | 1 year
  Cost-effectiveness, cost-utility and cost-benefit methods.

CONTACTS AND LOCATIONS:
Overall Officials: Roar Johnsen, phd prof, Study Director — Norwegian University of Science and Technology
Locations (2):
- Norway (2):
  - Hysnes Rehabilitation Centre, Rissa
  - St. Olavs University Hospital, Trondheim

REFERENCES:
- [Background] Fimland MS, Vasseljen O, Gismervik S, Rise MB, Halsteinli V, Jacobsen HB, Borchgrevink PC, Tenggren H, Johnsen R. Occupational rehabilitation programs for musculoskeletal pain and common mental health disorders: study protocol of a randomized controlled trial. BMC Public Health. 2014 Apr 16;14:368. doi: 10.1186/1471-2458-14-368. PMID 24735616
- [Result] Aasdahl L, Pape K, Vasseljen O, Johnsen R, Gismervik S, Halsteinli V, Fleten N, Nielsen CV, Fimland MS. Effect of Inpatient Multicomponent Occupational Rehabilitation Versus Less Comprehensive Outpatient Rehabilitation on Sickness Absence in Persons with Musculoskeletal- or Mental Health Disorders: A Randomized Clinical Trial. J Occup Rehabil. 2018 Mar;28(1):170-179. doi: 10.1007/s10926-017-9708-z. PMID 28401441
- [Result] Nordstoga AL, Mork PJ, Steiro Fimland M. Improved cardiorespiratory fitness after occupational rehabilitation in merged diagnostic groups. Ann Occup Environ Med. 2018 Feb 28;30:16. doi: 10.1186/s40557-018-0227-y. eCollection 2018. PMID 29507732
- [Result] Aasdahl L, Pape K, Vasseljen O, Johnsen R, Fimland MS. Improved Expectations About Length of Sick Leave During Occupational Rehabilitation Is Associated with Increased Work Participation. J Occup Rehabil. 2019 Sep;29(3):475-482. doi: 10.1007/s10926-018-9808-4. PMID 30151631
- [Result] Aasdahl L, Pape K, Vasseljen O, Johnsen R, Gismervik S, Jensen C, Fimland MS. Effects of Inpatient Multicomponent Occupational Rehabilitation versus Less Comprehensive Outpatient Rehabilitation on Somatic and Mental Health: Secondary Outcomes of a Randomized Clinical Trial. J Occup Rehabil. 2017 Sep;27(3):456-466. doi: 10.1007/s10926-016-9679-5. PMID 27815771
- [Result] Skagseth M, Fimland MS, Ivar Lund Nilsen T, Aasdahl L. Physical activity after inpatient occupational rehabilitation: Secondary outcomes of two randomized controlled trials. Scand J Med Sci Sports. 2020 Feb;30(2):339-348. doi: 10.1111/sms.13577. Epub 2019 Oct 30. PMID 31609021